CLINICAL TRIAL: NCT00001448
Title: The Effect of Oral Candidiasis on the Speech Production, Feeding Skills, and Self-Concept of Children and Adolescents With Symptomatic HIV Infection
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950185; 95-C-0185
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-07

CONDITIONS: Candidiasis, Oral; Eating Disorders; HIV Infections; Speech Disorders
Keywords: Antifungal Therapy; Articulation; Behavior; Expressive Language; Thrush
MeSH Terms: conditions — Candidiasis, Oral; Feeding and Eating Disorders; HIV Infections; Speech Disorders; Behavior

SUMMARY:
The main objectives of this study are: 1) to determine whether various levels of severity of oral candidiasis (thrush) in the child are associated with different levels of speech production, feeding skills, and self-concept, and 2) to assess the effect of the reduction of oral thrush over time on the speech function, feeding skills, and self-concept in HIV-infected patients who already are receiving various antifungal medications for treatment of their thrush (Note: Decisions regarding antifungal therapy are made completely independent from this study).

Children with HIV disease, ages 6-21 years, who have oral thrush are eligible to paricipate in the study. The child and his/her parent will be asked to complete a variety of measures at specific time intervals over approximately one month during visits to the National Institutes of Health for treatment on other protocols. First, a nurse will rate the location and severity of thrush in the child's mouth. Then the parent will complete questionnaires assessing the effect of oral thrush on the child's feeding and speech skills and everyday functioning. Finally, the child will be administered a brief speech and oral-motor evaluation and will complete some questionnaires about how the thrush affects his/her day-to-day activities and self-concept.

The results of this study may help to better understand the cause of expressive language deficits observed in some children with HIV infection. More specifically, it will determine if any speech and feeding problems of HIV-infected children are associated with oral thrush. Learning more about the impact of oral thrush on the speech, feeding, and the self-concept of children with HIV disease may be used for parent and patient education and to develop rehabilitative recommendations to benefit HIV-infected patients with oral thrush.

DETAILED DESCRIPTION:
Language impairments in children with symptomatic HIV infection are associated with the direct effects of HIV on the central nervous system (CNS). Furthermore, expressive language is more vulnerable to the effects of HIV compared to receptive language (Wolters, et al., 1995). Several factors, however, are likely to be involved in producing the expressive language impairments observed in the HIV-infected pediatric population. Oral candidiasis (thrush), a fungal infection in the oral cavity that frequently appears in HIV-infected children (Walsh, 1994), also may contribute to speech and language deficits depending on the severity of the thrush. Feeding skills and self-concept may be negatively affected by oral thrush as well.

The effect of oral candidiasis on the speech production, feeding skills, and self-concept of children and adolescents with HIV infection will be examined in this pilot study. Several disciplines (Neuropsychology, Speech, Nursing, and Infectious Disease) will be involved to investigate the severity of oral candidiasis on various aspects of everyday behavior.

Interdisciplinary assessment of the ramifications of oral thrush on speech production and feeding skills have not been conducted to date in children or adolescents infected with HIV. Most studies have assessed only single dimensions or functions such as language or they have yielded only descriptive data, for example, regarding the severity of oral thrush. This pilot study, however, will investigate the association between oral thrush and speech and feeding dysfunction using some newly-developed measures. The study will also examine whether oral candidiasis may influence the self-concept of children and adolescents with HIV infection.

ELIGIBILITY:
Children and adolescents with HIV infection, ages 6 through 21 years of age, who are treated in other protocols at the Pediatric Branch of the National Cancer Institute (NCI) and have oral candidiasis as determined by the Pediatric Nurse Practitioners, are eligible to participate in this study.

Children and adolescents with infections or diseases other than candidiasis affecting the oral cavity as determined by the PNP's during the physical exam will be excluded from the study.

Furthermore, patients who are identified by the speech pathologist to have oro-facial structural and/or functional abnormalities that cause a significant disturbance in speech, voice, or swallowing will be excluded.

Children will also not be able t participate in the study if they cannot understand the measures, even if the questions are read to them, which will be determined by the Neuropsychology staff.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1995-08; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Epstein LG, Sharer LR, Oleske JM, Connor EM, Goudsmit J, Bagdon L, Robert-Guroff M, Koenigsberger MR. Neurologic manifestations of human immunodeficiency virus infection in children. Pediatrics. 1986 Oct;78(4):678-87. PMID 2429248
- [Background] Pressman H. Communication disorders and dysphagia in pediatric AIDS. ASHA. 1992 Jan;34(1):45-7. No abstract available. PMID 1540256
- [Background] Wolters PL, Brouwers P, Moss HA, Pizzo PA. Differential receptive and expressive language functioning of children with symptomatic HIV disease and relation to CT scan brain abnormalities. Pediatrics. 1995 Jan;95(1):112-9. PMID 7770287